CLINICAL TRIAL: NCT01022125
Title: A Phase I Study in Healthy Subjects to Assess the Relative Bioavailability of TMC435 Following Administration of Potential Phase III Formulations Compared to the Phase IIb Capsule and to Assess the Effect of Food on the Bioavailability of TMC435 Following Intake of the Phase IIb Capsule
Brief Title: TMC435-TiDP16-C121: A Study Comparing 2 Tablet Formulations of TMC435 to an Established Capsule Formulation and Evaluating the Effect of Food on Blood Levels of TMC435
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Compound Development Team Leader, Tibotec Pharmaceuticals, Ireland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR016744
Record Dates: First submitted 2009-11-25; First posted 2009-12-01 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-05

CONDITIONS: Hepatitis C Virus
Keywords: TMC435-TiDP16-C121; TMC435-C121; TMC435; TMC435350; Protease inhibitor; HCV; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir

INTERVENTIONS:
Drug: TMC435

SUMMARY:
The purpose of this study is to compare the levels of TMC435 in the blood circulation after intake of 2 tablet formulations with the level of TMC435 in the blood circulation after intake of a capsule formulation. The trial will also evaluate levels of TMC435 in the blood circulation after intake of the capsule formulation fasted or following a meal.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), open-label (all people involved know the identity of the intervention), single dose, crossover (volunteers will receive different interventions sequentially during the trial) study in healthy volunteers. The trial will evaluate the levels of TMC435 in the blood circulation after a single dose of 150 mg TMC435 as a capsule formulation taken fasted (Treatment A) and following a meal (Treatment B). In addition, the study will evaluate the levels of TMC435 in the blood circulation after intake of a single dose of 150 mg TMC435 as 2 different tablet formulations (Treatments C and D). There will be a 14-day washout period between treatments and a 4-5 week follow-up at the end. Each volunteer will receive all four treatments. The main focus of the trial is the pharmacokinetic characteristics (how drugs are absorbed in the body, how they are distributed within the body and how they are removed from the body over time) of the different formulations. This evaluation requires multiple blood samples from Day 1 through 72 hours after dosing. Safety assessments (lab work, blood pressure, pulse and electrocardiogram) will follow a different schedule and are measured on Day -1 (day prior to taking first dose of drug), Day 1 (day of first dosing) and/or Day 4 of each treatment period, and 4 weeks after the last treatment. Each volunteer will receive 4 treatments, about 14 days apart from each other. Each treatment consists of one single dose of 150 mg TMC435.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker for at least 3 months
* Body Mass Index of 18.0 to 30.0 kg/m2
* Healthy based on a medical evaluation including medical history, physical examination, blood tests and electrocardiogram

Exclusion Criteria:

* Infection with Hepatitis A, B or C virus
* Infection with the human immunodeficiency virus (HIV)
* Women who are pregnant or breastfeeding
* History of, or any current medical condition which could impact the safety of the participant in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Rate and extent of absorption of TMC435 following administration of the tablet vs the capsule formulations and rate and extent of absorption of TMC435 following administration of the capsule formulation fasted or with food | Measured over a period of 4 consecutive days (Day1-Day4) per treatment. Treatments (4) are 14 days apart from each other. During 1st day of each treatment, 10 blood samples for determination of pharmacokinetic characteristics are taken.

SECONDARY OUTCOMES:
Safety and tolerability following administration of single doses of 150 mg TMC435 | AEs: continuously: laboratory, vital signs and ECG parameters: 3 visits per treatment, for 4 treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited